CLINICAL TRIAL: NCT03719508
Title: Predictive Value of Various Nutritional Screening and Assesment Tools and a Surgery Scoring System (POSSUM Score) for Predicting Postoperative Complications in Patients Scheduled for Abdominal Surgery
Brief Title: Preoperative Nutritional Assessment for Predicting Complications Risk in Patients Undergoing Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Dimitrios Karayiannis, Clinical Dietitian, Department of Clinical Nutrition and Metabolism, Evangelismos Hospital
Other Study IDs: 23/27-01-2014
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Abdominal Surgery
Keywords: Nutritional assesment; Nutritional screening tools; Abdominal Surgery; Stomach Neoplasms; Colorectal Surgery
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Predictive Value of Various Nutritional Screening and Assesment Tools and a Surgery Scoring System (POSSUM Score) for Predicting Postoperative Complications in Patients Scheduled for Abdominal Surgery.

DETAILED DESCRIPTION:
Preoperative malnutrition in surgical patients is an established risk factor of peri-operative morbidity and mortality, post-operative complications, infections and increased length of hospital stay. The reported prevalence of malnutrition in gastrointestinal (GI) and major abdominal surgery patients ranges from 30% to 50%. For these reasons it is important to recognize malnourished patients before surgery in order to provide the most appropriate preoperative nutritional therapy which will in turn improve nutritional status and reduce postoperative complications and length of hospital stay.

The aim of the present study was to compare the prognostic power of different screening tools for post - op complications. This was a prospective observational cohort study, performed in patients scheduled for an abdominal operation in the Second Department of Surgery, Evangelismos General Hospital in Athens, Greece. All patients were screened at admission and before operation. Data were collected in a special form by the dietician and the surgeon, with the use of screening tools and the local Electronic Medical Record System called "Emrora". Patients were followed up after surgery until discharge by the surgeon who recorded any complication or case of death in a new form.

ELIGIBILITY:
Inclusion Criteria:

* 18 years at least
* Diseases of the digestive tract (oesophageal, gastric or intestinal), or other abdominal diseases requiring elective surgery,

Exclusion Criteria:

* Age < 18
* Pregnancy
* Major coagulopathy
* Permanent pacemaker
* Specific preoperative nutritional support before admission to hospital
* Unable to give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged at least 18 years who presented with diseases of the digestive tract (oesophageal, gastric or intestinal), or with other abdominal diseases requiring elective surgery.
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2013-01-05 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Postoperative clinical complications. | 3 months
  Number of respiratory, cardiovascular, renal, neurological, infectious and surgical after surgery. Complication will be defined by the Clavien-Dindo classification and our primary outcome will be long-term complications higher than grade III.

SECONDARY OUTCOMES:
Length of stay in hospital | 3 months
  Length of stay
All-cause mortality | 3 months
  All-cause mortality is assessed during in-hospital stay and 90 days after the date of surgery
Readmission | 6 months
  Readmission to the center within 180 days of the original procedure.
Accuracy of the POSSUM Scoring Systems to predict clinical complications and mortality. | 1 month
  Area Under the Receiver Operating Curve (ROC) as a Measure of the Accuracy of the P-POSSUM Scoring Systems to Predict clinical complications and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: George Stylianides, MD, PhD, Study Director — 2nd Department of Surgery
Locations (1):
- Department of Nutrition and Dietetics, Evaggelismos Hospital, Athens, Kolonaki, Greece

IPD SHARING:
Plan to Share IPD: No